CLINICAL TRIAL: NCT06749977
Title: Efficacy of Self-assembling Peptide P11-4 for the Treatment of Orthodontically Induced Initial Carious Lesions: a Randomized Clinical Trial
Brief Title: P11-4 and Fluoride Varnish for Remineralization of Post-orthodontic Lesions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Sofia (Other)
Responsible Party: Principal Investigator, Alexander Bonchev, Chief Assistant Professor Dr Alexander Bonchev, DMD, PhD, Medical University of Sofia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 76/ 8717
Record Dates: First submitted 2024-12-08; First posted 2024-12-27 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: White Spot Lesions
Keywords: white spot; SAP11-4; fluoride varnish; QLF
MeSH Terms: interventions — splicing factor 3a

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Treatment of WSL with SAP11-4 (Experimental): WSL were treated with SAP11-4 corresponding to the manufacturer's instructions.
  Interventions: Drug: Remineralization with SAP11-4
- Treatment of WSL with sodium fluoride varnish (Experimental): WSL were treated with sodium fluoride varnish corresponding to the manufacturer's instructions.
  Interventions: Drug: Remineralization with sodium fluoride varnish
- No treatment (No Intervention): No treatment

INTERVENTIONS:
Drug: Remineralization with SAP11-4 — The WSL were treated with SAP11-4 according to the manufacturer's instruction
  Arms: Treatment of WSL with SAP11-4
Drug: Remineralization with sodium fluoride varnish — The WSL were treated with sodium fluoride varnish according to the manufacturer's instruction
  Arms: Treatment of WSL with sodium fluoride varnish

SUMMARY:
This clinical study aims to compare the remineralizing effects of self-assembling peptide P11-4 (SAP11-4) with fluoride varnish in the treatment of post-orthodontic non-cavitated carious lesions (NCLs). The study uses the QLF camera to assess changes in lesion size, severity, and mineralization, evaluating the effectiveness of SAP11-4 in comparison to fluoride varnish or no treatment. The primary endpoint is the change in QLF parameters, alongside ICDAS scores and Nyvad criteria for clinical evaluation.

DETAILED DESCRIPTION:
NCLs are common after orthodontic treatment and can persist as white spot lesions, presenting an aesthetic concern. Fluoride is a standard treatment, but it primarily benefits the outer enamel surface, while SAP11-4 may potentially enhance remineralization within the lesion body by mimicking enamel matrix proteins. This clinical study seeks to compare the effectiveness of two treatments for post-orthodontic non-cavitated carious lesions (NCLs): self-assembling peptide P11-4 (SAP11-4) and fluoride varnish. The goal is to evaluate which treatment is more effective at promoting remineralization of these lesions. The study utilizes the Quantitative Light-induced Fluorescence (QLF) camera to monitor changes in lesion size, severity, and mineralization. This method allows for a detailed assessment of the effectiveness of SAP11-4 compared to fluoride varnish or no treatment at all. The primary outcome of the study is the change in QLF parameters, which will be measured alongside the International Caries Detection and Assessment System (ICDAS) scores and the Nyvad criteria, providing a comprehensive clinical evaluation of the treatments' effects on the carious lesions.

ELIGIBILITY:
Inclusion Criteria:

* - Patients (18-30 y old) with ≥ 20 permanent teeth were included in the study.
* Presence of non-cavitated accessible carious enamel lesions on the vestibular surfaces (ICDAS II codes 1 and 2) after debonding of the fixed orthodontic appliances that do not require invasive treatment.
* The patients completed the fixed orthodontic therapy within the past 2 weeks [48].
* No professional topical fluoride application during the last 6 months prior the study.
* Patients are able and voluntarily attend the study visits and have a proper oral hygiene during the study.
* A written informed consent was signed before the start of the study.
* Female patients declare no pregnancy and breast feeding.
* Stimulated salivary flow rate ≥ 1 ml/min.
* The patients have lived in the same geographic region with constant fluoride concentration in the water during the last five years.

Exclusion Criteria:

* - Previously treated NCLs.
* Teeth with carious lesions placed apart from the fixed orthodontic appliances.
* Presence of restorations in contact with the carious lesion.
* Previous application of remineralizing agent <6 months prior to study treatment.
* Evidence of tooth erosion.
* Patients with dental fluorosis, enamel hypoplasia or tetracycline pigmentation.
* Present health conditions like diabetes, history of head and neck illnesses, metabolic disorders affecting bone turnover.
* Immunosuppression drugs.
* Pregnant and breast-feeding women.
* Significantly reduced salivation (unstimulated/stimulated); concomitant medication intake, affecting salivary flow.
* Concurrent participation in another clinical trial.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2023-02-20 (Actual)

PRIMARY OUTCOMES:
QLF measuerement of the lesion's depth | Day 0, Day 120, Day 360
  The depth of the lesion (parameter deltaF) was monitored throughout the study period.
QLF measurement of the lesion's volume | Day 0, Day 120, Day 360
  The volume of the white spot lesion (parameter deltaQ) was monitored throughout the study period.
QLF measurement of the lesion's Area | Day 0, Day 120, Day 360
  The size of the white spot lesion (parameter Area) was monitored throughout the study period.

SECONDARY OUTCOMES:
International Caries Detection and Assessment System (ICDAS) score changes | Day 0, Day 120, Day 360
  The changes of the white spot lesion score of the ICDAS system were monitored throughout of the study period.
Caries activity assesment | Day 0, Day 120, Day 360
  The cnahges of the caries activity were monitored by the Nyvad criteria changes during the study period.

CONTACTS AND LOCATIONS:
Overall Officials: Radosveta I Vasileva, Clinical Professor, Study Chair — Medical University, Sofia; Alexander B Bonchev, Chief Assistant Professor, Principal Investigator — Medical University, Sofia
Locations (1):
- Medical University Sofia, Sofia, Bulgaria

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol
Time Frame: Starting in January 2025 till June 2025
Access Criteria: The access is generally limited to individuals and organizations involved in the study, as well as other authorized researchers, under specific conditions ensuring privacy and ethical use, controlled by the researchers of the particular study.